CLINICAL TRIAL: NCT02385214
Title: A Phase III, Multi-centre, Multi-national Randomised Control Trial Investigating 1cm v 2cm Wide Excision Margins for Primary Cutaneous Melanoma
Brief Title: MelmarT Melanoma Margins Trial Investigating 1cm v 2cm Wide Excision Margins for Primary Cutaneous Melanoma
Acronym: MelMarT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03.12; NCT01457157 (obsolete NCT alias)
Record Dates: First submitted 2014-06-13; First posted 2015-03-11 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cutaneous Melanoma by AJCC V7 Stage
Keywords: Malignant; Melanoma; Cancer; Surgery
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A Wide Local Excision = 1cm Margin (Experimental): ARM A: Experimental Arm Wide Local Excision = 1cm Margin + Sentinel Lymph Node Biopsy
  +/- Reconstruction
  Interventions: Procedure: Wide Local Excision = 1cm Margin
- Arm B Wide Local Excision = 2cm Margin (Active Comparator): ARM B:Control Arm Wide Local Excision = 2cm Margin + Sentinel Lymph Node Biopsy
  +/- Reconstruction
  Interventions: Procedure: Wide Local Excision = 2cm Margin

INTERVENTIONS:
Procedure: Wide Local Excision = 1cm Margin — A wide local excision involves removing an extra "safety margin" of healthy skin surrounding the original melanoma site to ensure that any remaining scattered melanoma tumour cells are removed that may have been left behind after the first initial biopsy/surgery.
  Arms: Arm A Wide Local Excision = 1cm Margin
Procedure: Wide Local Excision = 2cm Margin — A wide local excision involves removing an extra "safety margin" of healthy skin surrounding the original melanoma site to ensure that any remaining scattered melanoma tumour cells are removed that may have been left behind after the first initial biopsy/surgery.
  Arms: Arm B Wide Local Excision = 2cm Margin

SUMMARY:
Patients with a primary invasive melanoma are recommended to undergo excision of the primary lesion with a wide margin. There is evidence that less radical margins of excision may be just as safe. This is a randomised controlled trial of 1 cm versus 2 cm margin of excision of the primary lesion for adult patients with a primary invasive cutaneous melanomas >=1mm thick to determine differences in the rate of local recurrence and melanoma specific survival. A reduction in margins is expected to improve quality of life in patients

DETAILED DESCRIPTION:
This study will determine whether there is a difference in local recurrence rates and melanoma survival rates for patients treated with either a 1cm excision margin or 2cm margin for both intermediate & high risk melanomas. The study is designed to be able to prove or disprove that there is no difference in risk of the tumour recurring around the scar or anywhere else in the body between the two groups of patients. This study is designed to show that the risk of long-term pain associated with surgery can be halved. If the study shows no risk of the tumour recurrence then we will also be able to determine how much of an impact the narrower excision has on patients in terms of improved quality of life and reduced side effects from the surgery and melanoma disease. This trial will also evaluate and determine the economic impact of narrower excision margins on the health services and society in general.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a primary invasive cutaneous melanoma of Breslow thickness greater than 1 millimetre as determined by diagnostic biopsy (narrow excision, incision or punch biopsy) and subsequent histopathological analysis.
2. Patients must have had the invasive primary completely excised, including any in situ component but excluding melanocytic atypia, with a narrow margin, either in one stage or more than one stage in the case where an incision or punch biopsy has previously been performed. This information, including measured margins of lateral and deep clearance must be documented on the pathology report.
3. Must have a primary melanoma that is cutaneous (including head, neck, trunk, extremity, scalp, palm, sole).
4. An uninterrupted 2cm margin must be technically feasible around biopsy scar or primary melanoma.
5. Randomisation and the primary study intervention, including staging sentinel node biopsy, must be completed by 120 days of original diagnosis.
6. Patients must be 18 years or older at time of consent.
7. Patient must be able to give informed consent and comply with the treatment protocol and follow-up plan.
8. Life expectancy of at least 10 years from the time of diagnosis, not considering the melanoma in question, as determined by the PI.
9. Patients must have an ECOG performance score between 0 and 1.
10. A survivor of prior cancer is eligible provided that ALL of the following criteria are met and documented:

    * The patient has undergone potentially curative therapy for all prior malignancies,
    * There has been no evidence of recurrence of any prior malignancies for at least FIVE years (except for successfully treated cervical or non-melanoma skin cancer with no evidence of recurrence), and
    * The patient is deemed by their treating physician to be at low risk of recurrence from previous malignancies.

Exclusion Criteria:

1. Uncertain diagnosis of melanoma i.e. so-called 'melanocytic lesion of unknown malignant potential'.
2. Patient has already undergone wide local excision at the site of the primary index lesion.
3. Patient unable or ineligible to undergo staging sentinel lymph node biopsy of the primary index lesion.
4. Desmoplastic or neurotropic melanoma.
5. Microsatellitosis as per AJCC 2009 definition
6. Subungual melanoma
7. Patient has already undergone a local flap reconstruction of the defect after excision of the primary and determination of an accurate excision margin is impossible.
8. History of previous or concurrent (i.e., second primary) invasive melanoma.
9. Melanoma located distal to the metacarpophalangeal joint, on the tip of the nose, the eyelids or on the ear, mucous membranes or internal viscera.
10. Physical, clinical, radiographic or pathologic evidence of satellite, in-transit, regional, or distant metastatic melanoma.
11. Patient has undergone surgery on a separate occasion to clear the lymph nodes of the probable draining lymphatic field, including sentinel lymph node biopsy, of the index melanoma.
12. Any additional solid tumour or hematologic malignancy during the past 5 years except T1 skin lesions of squamous cell carcinoma, basal cell carcinoma, or uterine/cervical cancer.
13. Melanoma-related operative procedures not corresponding to criteria described in the protocol.
14. Planned adjuvant radiotherapy to the primary melanoma site after Wide Local Excision is not permitted as part of the protocol and any patients given this treatment would be excluded from the study.
15. History of organ transplantation.
16. Oral or parenteral immunosuppressive agents (not topical or inhaled steroids) at any time during study participation or within 6 months prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2015-01-03 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Local Melanoma Recurrence (Melanoma Specific Survival) | 0-120 months
  Time from randomisation to clinically, histologically or radiologically confirmed local recurrence of melanoma including satellite lesions and in transit metastases to regional draining lymph nodes.

SECONDARY OUTCOMES:
Recurrence-Free Survival | 0-120 months
  Time from randomisation to any clinical, histological or radiologically confirmed melanoma recurrence or death from any cause.
QoL and neuropathic pain assessments Neuropathic Pain (PainDetect) | Baseline, 3, 6 12, 24 & 60 months.
  Quality of Life
Overall Survival | 0-120 Months
  Time from randomisation to death from any cause.
Adverse events | Within 1 year
  An Adverse Event (AE) is any untoward medical occurrence in a participant administered a treatment which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavourable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the treatment timing, whether or not considered related to the treatment. An AE is any adverse change (developing or worsening) from the participant's pre-treatment condition, including intercurrent illness.
  AEs and any pre-existing medical conditions will be recorded at the Baseline assessment and routinely at Follow Up, until the participant completes the study, withdraws or dies.
Surgery related adverse events | Up to 30 days from randomisation
  The following surgical adverse events will be recorded from the time of trial treatment to 30 days following the wide excision (inclusive):
  * wound separation
  * seroma/haematoma at wide local excision site
  * haemorrhage
  * infection
  * skin graft failure
  * necrosis of flap used for reconstruction
  * deep venous thrombosis
  * urinary tract infection
  * pneumonia
  * cardiac complications
Health System Resource Use | Baseline, 3, 6, 12, 24 and 60 months
  All hospitalisations and other interventions will be captured in order to measure resource use.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moncrieff, Principal Investigator — Norfolk & Norwich University Hospital; Michael Henderson, Principal Investigator — Peter MacCallum Cancer Center
Locations (20):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States
- Australia (4):
  - Melanoma Institute Australia - Poche Centre, North Sydney, New South Wales
  - Gold Coast Melanom Clinic, Coolangatta, Queensland
  - Peter MacCallum Cancer Centre Division of Cancer Surgery, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Sunnybrook Health Sciences Centre, Toronto, Canada
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (13):
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, England
  - Guy's and St Thomas' Hospital NHS Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Mid Essex Hospital Services NHS Trust, Broomfield, Essex
  - St Helens & Knowsley NHS Trust, St Helens, Mersyside
  - Oxford University Hospitals NHS Trust, Headington, Oxford
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - St. James University Hospital, Leeds
  - Royal Free London NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Norfolk and Norwich University Hospital, Norwich

REFERENCES:
- [Derived] Temple-Oberle C, Nicholas C, Rojas-Garcia P. Current Controversies in Melanoma Treatment. Plast Reconstr Surg. 2023 Mar 1;151(3):495e-505e. doi: 10.1097/PRS.0000000000009936. Epub 2023 Feb 23. PMID 36821575
- See also: MASC Trials-Closed to recruitment page — https://www.masc.org.au/active-trials-closed-for-recruitment/